CLINICAL TRIAL: NCT00497939
Title: The Effectiveness of Saw Palmetto and Sanmiaoshan on International Prostate Symptom Score and Peak Urinary Flow Rate of Chinese Patients With Benign Prostatic Hyperplasia
Brief Title: The Effectiveness of Saw Palmetto and Sanmiaoshan on Benign Prostatic Hyperplasia in Chinese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2005.310-T; HARECCTR0500050
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Prostatic Hyperplasia; Adrenergic Alpha-Antagonists
Keywords: Benign Prostatic Hyperplasia (BPH); Currently on alpha blocker
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — saw palmetto extract

INTERVENTIONS:
Drug: Saw palmetto and sanmiaoshan capsule

SUMMARY:
The purpose of this study is to assess the effect of saw palmetto and sanmiaoshan, on top of alpha blocker, on urinary flow rate and BPH symptoms in patients with BPH.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 80 years old
* Clinically diagnosed to have BPH:

  * Suffered from lower urinary tract symptoms with IPSS>=8
  * Detectable prostatic enlargement determined by DRE
  * Urinary flow between 5 and 15ml/second in a total void volume >=150mL
  * Serum PSA level less than 4ng/ml or in between 4-10 ng/ml with percent free PSA >25% or>=4 with cancer excluded by biopsy

Exclusion Criteria:

* Acute retention of urine
* Congestive heart failure, unstable angina, arrhythmia, myocardial infraction
* Prostatic surgery
* Prostatic malignancy
* Gastrointestinal disease
* Renal impairment with serum creatinine >140 umol/l
* Hepatic disorder

Ages: 50 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-01; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Differences in IPSS between the study medication and placebo groups | At study enrolment, after six month of study medication or placebo administration, at the end of washout period and after six month of alternative drug treatment
Differences in Qmax between the study medication and placebo groups | At study enrolment, after six month of study medication or placebo administration, at the end of washout period and after six month of alternative drug treatment

SECONDARY OUTCOMES:
Differences in IPSS and Qmax at baseline and at the end of treatment drug / placebo treatment | From study enrolment/ after washout period to the end of study medication / placebo administration
Mean urinary flow rate, post-void residual volume, prostate volume, PSA and GHQ score between study medication group and placebo group | At study enrolment, after six month of study medication or placebo administration, at the end of washout period and after six month of alternative drug treatment
Mean urinary flow rate, post-void residual volume, prostate volume, PSA and GHQ score between study medication group and baseline, and placebo group and baseline | From study enrolment/ after washout period to the end of study medication / placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, Dr, Principal Investigator — Department of Surgery, Division of Urology, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China